CLINICAL TRIAL: NCT04324853
Title: Assessing the Effect of Maternal Helminth Infection on Vitamin D Regulation and on the Immune System of the Infant
Brief Title: Helminth Infection During Pregnancy on Vitamin D Regulation: HELMVIT Study
Acronym: HELMVIT
Status: Completed | Type: Observational
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Collaborators: Technical University of Munich (Other); University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: PROT N°038/2018/SG/CNE
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-04

CONDITIONS: Vitamin D Deficiency; Immunosuppression
Keywords: Pregnancy; Vitamin D; Helminth; Schistosomiasis
MeSH Terms: conditions — Vitamin D Deficiency; Schistosomiasis | interventions — Microscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — S. haematobium will be assessed using urine filtration technique, intestinal parasites will be determined using the Kato-Katz method as well as different culture methods
  According to their infection status, women will be allocated to the following groups: S. haematobium positive, geohelminths positive and helminth negative participants.
  Plasma and peripheral blood mononuclear cells (PBMCs) are prepared and stored at -150°C; serum will be collected and immediately frozen in lightproof vials at -80 °C until further analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- S. haematobium positive: Pregnant women infected with Schistosoma hematobium alone
  Interventions: Diagnostic Test: Microscopy ( Urine filtration), UCAA test, qPCR,
- geohelminths positive: pregnant women infected with geohelminths alone
  Interventions: Diagnostic Test: Microscopy (Kato Katz, Coproculture, Harada Mori, MIF), qPCR,
- Helminth negative: Pregnant women free of anyn helminths infection
  Interventions: Diagnostic Test: Microscopy (Kato Katz, Coproculture, Harada Mori, MIF), qPCR,

INTERVENTIONS:
Diagnostic Test: Microscopy ( Urine filtration), UCAA test, qPCR, — Schistosomiasis is an acute and chronic parasitic disease caused by blood flukes (trematode worms) of the genus Schistosoma.Schistosomiasis is prevalent in tropical and subtropical areas, especially in poor communities without access to safe drinking water and adequate sanitation.
  Groups: S. haematobium positive
Diagnostic Test: Microscopy (Kato Katz, Coproculture, Harada Mori, MIF), qPCR, — Soil-transmitted helminth infections are among the most common infections worldwide and affect the poorest and most deprived communities. They are transmitted by eggs present in human faeces which in turn contaminate soil in areas where sanitation is poor.
  Groups: Helminth negative; geohelminths positive

SUMMARY:
Purpose: To examine whether helminth infection during pregnancy alters Vitamin-D-metabolism and reactivity of the child's immune system

Hypothesis: Helminth infection during pregnancy is associated with altered Vitamin D levels and Vitamin D receptor expression in the placenta and modified immune reactivity in the infant.

DETAILED DESCRIPTION:
Objectives The primary objective of the proposed research project is to study the impact of helminth infection in general and particularly of infection with S. haematobium during pregnancy on Vitamin D metabolism and its related factors as well as the impact of maternal infection on infants developing immune system and health.

Specific Objectives To assess the effect of maternal helminths infections on Vitamin D and vitamin-D-related factors in the serum of pregnant women and cord blood of their infants,

To assess the effect of helminth infection on placental biology:

Determine expression levels of VDR and inflammatory genes Investigate histologically the gestational age and other functional aspects of the placenta Determine the influence of helminth driven inflammation and helminth antigens on placental tissue by establishing a (co-)culture system using primary placental cells and a placental cell line To assess whether helminth infections influence the infant's peripheral immune system by analyzing composition, reactivity and lineage determination of fetal cord blood mononuclear cells (CBMCs) in relation to the maternal and fetal immune and Vitamin D status.

Current study focusing objectives In the present study the investigators explore if and how Vitamin D and its related signals are modulated by helminth infection and how helminth infection could thereby shape the developing immune system of the newborn by analyzing CBMCs.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending antenatal care from Lambaréné and Fougamou areas
* Pregnant women who have given written informed consent to the study for herself and for her unborn child and live infant.

Exclusion Criteria:

* Known of chronic infections and diseases(e.g. diabetes, HIV, Hepatitis B and C, anemia).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target population is pregnant women coming to the ante natal clinics (ANC) for routine visits or to obtain medical care in the obstetrics department of the Albert Schweitzer Hospital (ASH) as well as at Georges Rawiri General Hospital (GRGH), both situated in Lambaréné. The pregnant women originally from areas endemic for Schistosomiasis and Soil-transmitted helminths will be invited to participate into the study.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Association between Schistosoma and helminth infection and Vitamin D levels. | 48 Months
  Schistosoma hematobium in pregnancy is associated with vitamin D metabolism

SECONDARY OUTCOMES:
Association between Schistosoma infection and intrauterine growth restriction (IUGR) (defined as birth weight below the 10th birth weight percentile), stillbirth and premature delivery. | 48 Months
  Schistosoma hematobium infection during pregnancy is associated with a birth weight born child

CONTACTS AND LOCATIONS:
Overall Officials: Ayola A ADEGNIKA, MD, PhD, Principal Investigator — Centre de Recherche Médicale de Lambaréné; Meral Esen, MD, Study Chair — University Hospital Tuebingen; Clarissa DaCosta, MD, Study Director — Technical University of Munich
Locations (1):
- Josiane Y Honkpehedji, Lambaréné, Moyen-Ogooué Province, Gabon